CLINICAL TRIAL: NCT02451774
Title: SAFETY AND EFFICACY OF PENTOXIFYLLINE VERSUS PLACEBO ADMINISTERED AS APOPTOSIS INDUCTOR DURING REMISSION INDUCTION PHASE OF PEDIATRIC PATIENTS WITH ACUTE LYMPHOBLASTIC LEUKEMIA
Brief Title: Pentoxifylline In Pediatric Acute Lymphoblastic Leukemia During Induction
Acronym: PTX-II
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramón Óscar González-Ramella, Ph.D (Other)
Collaborators: Instituto de Investigacion en Cancer de la Infancia y la Adolescencia (Unknown); Hospital Civil Juan I. Menchaca (Other); Centro de Investigacion Biomedica de Occidente (Unknown)
Responsible Party: Sponsor-Investigator, Ramón Óscar González-Ramella, Ph.D, PhD in immunology, University of Guadalajara
Organization: University of Guadalajara (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IICIA -PTX02
Record Dates: First submitted 2015-02-09; First posted 2015-05-22 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: pediatric; apoptosis
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Pentoxifylline; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pentoxifylline Plus Chemotherapy (Experimental): Pentoxifylline: 10-20 milligrams per kilogram, doses daily by oral, for 30 days.
  Chemotherapy: Prednisone, Vincristine, Daunorubicin, L-asparaginase, Cyclophosphamide, Cytarabine, 6-Mercaptopurine, Methotrexate, Hydrocortisone and Cytarabine
  Interventions: Drug: Pentoxifylline Plus Chemotherapy
- Placebo Plus Chemotherapy (Placebo Comparator): Placebo: double blind period, one doses daily for 30 days. Chemotherapy: Prednisone, Vincristine, Daunorubicin, L-asparaginase, Cyclophosphamide, Cytarabine, 6-Mercaptopurine, Methotrexate, Hydrocortisone and Cytarabine
  Interventions: Drug: Placebo Plus Chemotherapy

INTERVENTIONS:
Drug: Pentoxifylline Plus Chemotherapy — Pentoxifylline 10 to 20 milligrams per kilogram, daily, for up to 32 days Chemotherapy: Prednisone 40 milligrams per square meter per day, orally, day 5-32. Vincristine 1.5 milligrams per square meter per week, intravenously, day 5, 12, 19, 26. Daunorubicin 25 milligrams per square meter per week, intravenously, days 5; 12. L-asparaginase 10,000 units for square meter, intramuscular, days 6, 8, 10, 12, 14, 16, 19, 21, 23. Cyclophosphamide 1000 milligrams per square meter per dose intravenously, day 26. Cytarabine 75 milligrams per square meter per dose intravenously, days 27-30, 34-37. 6-Mercaptopurine 60 milligrams per square meter per dose, orally, days 26-39, Mix: Methotrexate 8-12 milligrams, Hydrocortisone 16-24 milligrams and Cytarabine 24-36 milligrams, intrathecal, day 19.
  Other Names: Oxpentifylline
  Arms: Pentoxifylline Plus Chemotherapy
Drug: Placebo Plus Chemotherapy — Placebo daily, for up to 32 days Chemotherapy: Prednisone 40 milligrams per square meter per day, orally, day 5-32. Vincristine 1.5 milligrams per square meter per week, intravenously, day 5, 12, 19, 26. Daunorubicin 25 milligrams per square meter per week, intravenously, days 5; 12. L-asparaginase 10,000 units for square meter, intramuscular, days 6, 8, 10, 12, 14, 16, 19, 21, 23. Cyclophosphamide 1000 milligrams per square meter per dose intravenously, day 26. Cytarabine 75 milligrams per square meter per dose intravenously, days 27-30, 34-37. 6-Mercaptopurine 60 milligrams per square meter per dose, orally, days 26-39, Mix: Methotrexate 8-12 milligrams, Hydrocortisone 16-24 milligrams and Cytarabine 24-36 milligrams, intrathecal, day 19.
  Other Names: Placebo
  Arms: Placebo Plus Chemotherapy

SUMMARY:
Recent advances in acute lymphoblastic leukemia treatment are based on a cytotoxic drug combination. Measurement of minimal residual disease in bone marrow samples at day 14 of treatment is the most powerful early predictive indicator of further relapse, and it can be applied practically to all patients with acute lymphoblastic leukemia. Even more so, it has been observed that patients who present negative minimal residual disease in bone marrow samples at day 7 during induction have a better prognosis than those achieving this at day 14.

Relapse represents the main cause of treatment failure that related in the extreme with resistance to apoptosis, defining the latter as the principal mechanism of programmed cell death; it is also related with the induction of leukemic cells to senescent arrest.

Pentoxifylline is a methyl-xanthine byproduct considered an unspecific inhibitor of phosphodiesterase. It inhibits nuclear factor-kappa-beta activation by different mechanisms and stimulates apoptosis induced by different drugs; thus, it can optimize the antineoplastic effect of actual treatments in order to increase the apoptosis of leukemic cells. This effect might improve the prognosis of these patients.

Evaluate the safety and effect of Pentoxifylline together with antineoplastic drugs in order to study increased apoptosis and decreased senescence during the remission induction phase in pediatric patients with newly diagnosed acute lymphoblastic leukemia. To achieve this propose, we will divide patients in two groups, who will receive pentoxifylline or placebo depending on the group, in addition to conventional treatment according to the protocol standard chemotherapy schema for pediatric patients with acute lymphoblastic leukemia at our institution during the remission induction phase. In addition, we will test whether the study group exerts an impact on reaching remission earlier as compared with the control group.

DETAILED DESCRIPTION:
This study will be controlled, double-blind clinical trial versus placebo, with random assignment to evaluate the effect of pentoxifylline on apoptosis and senescence of leukemic blasts from remission induction in pediatric patients with newly diagnosed acute lymphoblastic leukemia, as well as to address pentoxifylline efficacy and safety in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and teenaged patients of both genders ≤18 years of age with newly diagnosed acute lymphoblastic leukemia in accordance with French-American-British criteria and under immunophenotypical classification and paired within the risk-classification group.
* Patients with ≥20 kg of weight at the time of treatment assignment.
* Patients who are able to swallow the medicine
* Patients agreeing to enter the protocol by the signing of informed consent by the parent
* Patients who could give their assent to enter the protocol
* The parent or guardian must be able to read.

Exclusion Criteria:

* Patients with treatment adherence of ≥80 percent
* Patients or their parents who decide to abandon the study or who withdraw consent for participation
* Patients who present grade III or higher adverse event.
* Patients previously treated with chemotherapy and/or radiotherapy
* History of peptic acid disease or gastrointestinal bleeding
* Known pentoxifylline intolerance and general intolerance to xanthine, caffeine or theophylline
* Patients in treatment with anticoagulants, Cimetidine, Ciprofloxacin, or Theophylline
* Patients with Down syndrome
* Patients with several bleeding or extensive retinal hemorrhage, several cardiac arrhythmias (paroxysmal supraventricular tachycardia, congenital atrioventricular block, arrhythmias associated with congenital heart disease, digital poisoning, and patients after cardiac surgery, hypoxia, hypercapnia, and electrolyte disturbances)
* Patients with hypotension
* Several liver failures
* Bleeding diathesis (for bleeding disorders or anticoagulant medication)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Apoptosis measure by Flow Cytometry | Up to 28 days after initiation of chemotherapy for remission induction
  Percentage of apoptotic cells by Flow Cytometry

SECONDARY OUTCOMES:
Senescence measure by Flow Cytometry | Up to 28 days after initiation of chemotherapy for remission induction.
  Percentage of senescent blasts by Flow Cytometry
Safety measure by Common Terminology Criteria for Adverse Events version 4.0 | Evaluate frequency adverse events with pentoxifylline up to 6 weeks
  Percentage of adverse events grading table is a list of common terms and severity (intensity) of parameters used to describe adverse events occurring in Common Terminology Criteria for Adverse Events version 4.0

OTHER OUTCOMES:
Gene expression measure by Microarray and Semi-quantitative Polymerase Chain Reaction. | Up to 28 days after initiation of chemotherapy for remission induction.
  Fold change by microarray and Semi-quantitative Polymerase Chain Reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ramón O. Gonzalez Ramella, PhD, Principal Investigator — Instituto de Investigacion de Cancer de la Infancia y la Adolescencia
Locations (1):
- Hospital Civil de Guadalajara "Dr. Juan I. Menchaca", Guadalajara, Jalisco, Mexico

REFERENCES:
- [Result] Makishima H, Visconte V, Sakaguchi H, Jankowska AM, Abu Kar S, Jerez A, Przychodzen B, Bupathi M, Guinta K, Afable MG, Sekeres MA, Padgett RA, Tiu RV, Maciejewski JP. Mutations in the spliceosome machinery, a novel and ubiquitous pathway in leukemogenesis. Blood. 2012 Apr 5;119(14):3203-10. doi: 10.1182/blood-2011-12-399774. Epub 2012 Feb 9. PMID 22323480
- [Result] Dores GM, Devesa SS, Curtis RE, Linet MS, Morton LM. Acute leukemia incidence and patient survival among children and adults in the United States, 2001-2007. Blood. 2012 Jan 5;119(1):34-43. doi: 10.1182/blood-2011-04-347872. Epub 2011 Nov 15. PMID 22086414
- [Result] Perez-Saldivar ML, Fajardo-Gutierrez A, Bernaldez-Rios R, Martinez-Avalos A, Medina-Sanson A, Espinosa-Hernandez L, Flores-Chapa Jde D, Amador-Sanchez R, Penaloza-Gonzalez JG, Alvarez-Rodriguez FJ, Bolea-Murga V, Flores-Lujano J, Rodriguez-Zepeda Mdel C, Rivera-Luna R, Dorantes-Acosta EM, Jimenez-Hernandez E, Alvarado-Ibarra M, Velazquez-Avina MM, Torres-Nava JR, Duarte-Rodriguez DA, Paredes-Aguilera R, Del Campo-Martinez Mde L, Cardenas-Cardos R, Alamilla-Galicia PH, Bekker-Mendez VC, Ortega-Alvarez MC, Mejia-Arangure JM. Childhood acute leukemias are frequent in Mexico City: descriptive epidemiology. BMC Cancer. 2011 Aug 17;11:355. doi: 10.1186/1471-2407-11-355. PMID 21846410
- [Result] Belson M, Kingsley B, Holmes A. Risk factors for acute leukemia in children: a review. Environ Health Perspect. 2007 Jan;115(1):138-45. doi: 10.1289/ehp.9023. PMID 17366834
- [Result] Pui CH, Robison LL, Look AT. Acute lymphoblastic leukaemia. Lancet. 2008 Mar 22;371(9617):1030-43. doi: 10.1016/S0140-6736(08)60457-2. PMID 18358930
- [Result] Pui CH, Carroll WL, Meshinchi S, Arceci RJ. Biology, risk stratification, and therapy of pediatric acute leukemias: an update. J Clin Oncol. 2011 Feb 10;29(5):551-65. doi: 10.1200/JCO.2010.30.7405. Epub 2011 Jan 10. PMID 21220611
- [Result] Wong RS. Apoptosis in cancer: from pathogenesis to treatment. J Exp Clin Cancer Res. 2011 Sep 26;30(1):87. doi: 10.1186/1756-9966-30-87. PMID 21943236
- [Result] Herr I, Debatin KM. Cellular stress response and apoptosis in cancer therapy. Blood. 2001 Nov 1;98(9):2603-14. doi: 10.1182/blood.v98.9.2603. PMID 11675328
- [Result] Campisi J. Aging, cellular senescence, and cancer. Annu Rev Physiol. 2013;75:685-705. doi: 10.1146/annurev-physiol-030212-183653. Epub 2012 Nov 8. PMID 23140366
- [Result] Sankari SL, Masthan KM, Babu NA, Bhattacharjee T, Elumalai M. Apoptosis in cancer--an update. Asian Pac J Cancer Prev. 2012;13(10):4873-8. doi: 10.7314/apjcp.2012.13.10.4873. PMID 23244073
- [Result] Chauhan PS, Bhushan B, Singh LC, Mishra AK, Saluja S, Mittal V, Gupta DK, Kapur S. Expression of genes related to multiple drug resistance and apoptosis in acute leukemia: response to induction chemotherapy. Exp Mol Pathol. 2012 Feb;92(1):44-9. doi: 10.1016/j.yexmp.2011.09.004. Epub 2011 Oct 19. PMID 22037714
- [Result] Reuter S, Gupta SC, Kannappan R, Aggarwal BB. WITHDRAWN: Evidence for the critical roles of NF-kappaB p65 and specificity proteins in the apoptosis-inducing activity of proteasome inhibitors in leukemia cells. Biochim Biophys Acta. 2012 Jan 10:10.1016/j.bbadis.2012.01.002. doi: 10.1016/j.bbadis.2012.01.002. Online ahead of print. PMID 22265847
- [Result] Hernandez-Flores G, Ortiz-Lazareno PC, Lerma-Diaz JM, Dominguez-Rodriguez JR, Jave-Suarez LF, Aguilar-Lemarroy Adel C, de Celis-Carrillo R, del Toro-Arreola S, Castellanos-Esparza YC, Bravo-Cuellar A. Pentoxifylline sensitizes human cervical tumor cells to cisplatin-induced apoptosis by suppressing NF-kappa B and decreased cell senescence. BMC Cancer. 2011 Nov 10;11:483. doi: 10.1186/1471-2407-11-483. PMID 22074157
- [Result] Armstrong SA, Look AT. Molecular genetics of acute lymphoblastic leukemia. J Clin Oncol. 2005 Sep 10;23(26):6306-15. doi: 10.1200/JCO.2005.05.047. PMID 16155013
- [Derived] Salceda-Rivera V, Ortiz-Lazareno PC, Hernandez-Flores G, Vazquez-Urrutia JR, Meza-Arroyo J, Pardo-Zepeda M, Romo-Rubio H, Barba-Barba C, Sanchez-Zubieta F, Barron-Gallardo CA, Gonzalez-Ramella O, Bravo-Cuellar A. Very early remission and increased apoptosis with the use of Pentoxifylline in children with acute lymphoblastic leukemia. Front Oncol. 2024 Oct 3;14:1401262. doi: 10.3389/fonc.2024.1401262. eCollection 2024. PMID 39421449